CLINICAL TRIAL: NCT00811876
Title: Monitoring Tolerance, Safety and Acceptance of Depo-Eligard® in an Open Label, Retrospective, Non-interventional Clinical Trial
Brief Title: Retrospective, Non-interventional Study of Depo-Eligard®.
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Other Study IDs: BE-08-EGD-02
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data Collection on Depo-Eligard exposure — Retrospective, Non-interventional
  Other Names: leuproreline acetate exposure

SUMMARY:
Study will evaluate the real-world effectiveness of Depo-Eligard® after six months of treatment

DETAILED DESCRIPTION:
The study will provide data on the tolerance, safety and acceptance of Depo-Eligard® (leuproreline acetate) when used in routine clinical practice. Data on efficacy parameters such as testosterone, PSA levels, symptoms and treatment failure, if available will be collected.It will reflect the way Depo-Eligard® is used in routine clinical practice and how PSA, testosterone levels, symptoms and treatment failure, are used as parameters in the treatment for Prostate Cancer.

Patient data will be collected after a treatment period of six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients having been prescribed Depo-Eligard® in accordance with the terms of the marketing authorization
* Patients on treatment with Depo-Eligard® for at least six months
* Written consent has been obtained

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Belgian participating investigator sites having been prescribed Depo-Eligard® in accordance with the terms of the marketing authorization, on treatment with Depo-Eligard® for at least six months.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Tolerance, Safety (Adverse drug reactions, overall evaluation of safety and tolerability) and Acceptance of Depo-Eligard® | After at least 6 months treatment with Depo-Eligard

SECONDARY OUTCOMES:
Measurement of PSA and testosterone levels if available | After at least 6 months treatment with Depo-Eligard
Overall evaluation of efficacy | After a least 6 months treatment with Depo-Eligard
Overall patient assessment of treatment benefit | After at least 6 months treatment with Depo-Eligard

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (21):
- Belgium (21):
  - Antwerp
  - Berlaar
  - Bornem
  - Brussels
  - Charleroi
  - Ghent
  - Jemeppe
  - Kortrijk
  - Leuven
  - Liège
  - Lommel
  - Merksem
  - Mons
  - Mortsel
  - Ragnies
  - Tienen
  - Tongeren
  - Turnhout
  - Waregem
  - Willebroek
  - Yvoir